CLINICAL TRIAL: NCT06138925
Title: Analysis of the Psychometric Properties of Kinematic Parameters of Locomotion Measured by Inertial Measurement Units. Validation in Healthy Children and Children with Cerebral Palsy
Acronym: KAPP-IMU anc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ORNETTI 2023
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- healthy children (Active Comparator)
  Interventions: Other: Analysis of walking; Other: Analysis of running
- hildren with cerebral palsy (Experimental)
  Interventions: Other: Analysis of walking

INTERVENTIONS:
Other: Analysis of walking — 3-dimensional gait analysis with inertial measurement units (IMUs) on flat ground at different speeds (slow, comfortable and fast)
  Arms: healthy children
Other: Analysis of running — analysis of running on flat ground at different speeds (comfortable and fast)
  Arms: healthy children
Other: Analysis of walking — 3-dimensional gait analysis with inertial measurement units (IMUs) on flat ground at spontaneous speed (comfortable).
  Arms: hildren with cerebral palsy

SUMMARY:
Cerebral palsy (CP) is currently one of the major causes of disability in children. The presence of various disorders (muscle stiffness, architectural bone defects, spasticity) leads to a number of functional impacts, including severe impairment of mobility, particularly locomotion. Locomotion can be assessed using a motion capture system that enables 3-dimensional analysis, in order to help make treatment decisions and quantify them. Although these systems are currently considered to be the gold standard, the fact remains that they cause a certain amount of patient fatigue (long set-up times) and that walking is assessed in a laboratory rather than in real life.

Today, technological advances have brought to the fore other gait analysis devices, such as inertial measurement units (IMUs). Various systems incorporating IMUs in the feet, for example, respond to these problems of analysing walking in real-life situations. The IMUs record the movements and orientation of the foot in space; the data is then processed by algorithms to recognise walking steps and calculate the spatio-temporal parameters of locomotion. Additional IMUs positioned on the body can be grafted onto this system to provide a more precise analysis of locomotion, in particular by calculating the movements of the various joints of the lower limb. However, before such devices can be used in a pathological paediatric population, they must be validated in a healthy population. This validation must be conducted using a precise method that has been widely documented in the COSMIN recommendations (Consensus-based Standards for the selection of health Measurement Instruments). The first stage will assess the safety of the IMU devices in a healthy paediatric population, and the validity of the spatio-temporal parameters. If these properties are deemed to be compliant, these same parameters will be assessed in a paediatric population with cerebral palsy in the second stage.

ELIGIBILITY:
Inclusion Criteria:

* Children who have given their consent and whose legal representatives have given their consent
* Age between 7 and 17 years,
* Children able to understand simple commands and instructions.
* Children living within a maximum radius of 50 km of the investigation site.
* Child covered by national health insurance.

PATIENT GROUP (IN ADDITION TO THOSE ABOVE)

* Children with proven cerebral palsy resulting in locomotor impairment but able to move around without technical aids (cane, wheelchair).
* Child covered by national health insurance.

Exclusion Criteria:

* Children with a condition other than cerebral palsy that affects their ability to walk.
* Child subject to a measure of legal protection
* A child unable to give consent
* Pregnant, parturient or breast-feeding participant

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Walking speed | During the study visit
  participants' walking speed measured jointly by an IMU system in the shoe and a 3D locomotion analysis system

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No